CLINICAL TRIAL: NCT04866147
Title: Prediction Model Development for Chronic Postsurgical Pain in Adults
Brief Title: Prediction of Chronic Postsurgical Pain in Adults
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CPSP001122
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Chronic Postsurgical Pain; Acute Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Mastectomy, Segmental; Digestive System Surgical Procedures; Urogenital Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery patients: Patients who undergo various common surgical procedures
  Interventions: Procedure: Cardiothoracic surgery; Procedure: Breast surgery; Procedure: Gastrointestinal surgery; Procedure: Genitourinary surgery; Procedure: Orthopaedic surgery

INTERVENTIONS:
Procedure: Cardiothoracic surgery — Cardiac & large intrathoracic vessels, respiratory, thoracic, mediastinal & diaphragmatic procedures
Procedure: Breast surgery — Breast resections & mastectomies
Procedure: Gastrointestinal surgery — Digestive & spleen
Procedure: Genitourinary surgery — Urinary tract, genital & retroperitoneal tissue
Procedure: Orthopaedic surgery — Back & neck, shoulder & upper arm, hip & thigh, knees & lower leg

SUMMARY:
This research will be a prospective single-centre observational cohort study in Denmark spanning approximately one year. The objective of this study is to develop a clinically applicable and generalizable prediction model for postsurgical pain in adults.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Danish-speaking adults aged 18 years and older
* Patients who undergo common inpatient or outpatient surgical procedures

Exclusion Criteria:

* Patients with cognitive impairment
* Patients who refuse or unable to provide informed consent
* Patients who undergo re-operation within 3 months of their initial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergo surgery meeting inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1522 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Chronic post surgical pain | 3 months post surgery
  Pain related to the surgical procedure measured as average pain intensity on rest or movement using 11-point numeric rating scale (NRS; 0-10) where 0=no pain and 10=worst pain imaginable and/or average pain interference using 11-point NRS among any one of seven short-form Brief Pain Inventory items (general activity, mood, walking ability, normal work (including housework), relations with other people, sleep, enjoyment of life) in the past one week, where 0=pain does not interfere and 10=pain completely interferes.

SECONDARY OUTCOMES:
Acute post surgical pain | First 3 hours after surgery
  Acute post surgical pain intensity in the first 3 hours after surgery measured as pain at rest using 11-point numeric rating scale (NRS; 0-10) where 0=no pain and 10=worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, DMSc, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Silkeborg Regional Hospital, Silkeborg

REFERENCES:
- [Derived] Papadomanolakis-Pakis N, Haroutounian S, Sorensen JK, Runge C, Brix LD, Christiansen CF, Nikolajsen L. Development and internal validation of a clinical risk tool to predict chronic postsurgical pain in adults: a prospective multicentre cohort study. Pain. 2025 Mar 1;166(3):667-679. doi: 10.1097/j.pain.0000000000003405. Epub 2024 Sep 18. PMID 39297720